CLINICAL TRIAL: NCT03316482
Title: A Multicenter, Open, Prospective Study to Evaluate the Safety and Efficacy of Leuprorelin Acetate DPS (Leuplin DPS) Treatment Quarterly in Patients With Central Precocious Puberty
Brief Title: Leuprorelin Acetate DPS (Leuplin DPS) Treatment Quarterly in Patients With Central Precocious Puberty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jin Soon Hwang (Other)
Responsible Party: Sponsor-Investigator, Jin Soon Hwang, Professor, Ajou University School of Medicine
Organization: Ajou University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEUPLIN3M
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Leuprorelin treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leuplin DPS 11.25mg s.c. every 12 weeks (Experimental): Open
  Interventions: Drug: Leuplin DPS 11.25mg

INTERVENTIONS:
Drug: Leuplin DPS 11.25mg — Leuplin DPS 11.25mg s.c. every 12 weeks
  Other Names: injection

SUMMARY:
A multicenter, open-label, prospective study to evaluate the safety and efficacy of leuprorelin acetate DPS (Leuplin DPS) treatment quarterly in patients with central precocious puberty

DETAILED DESCRIPTION:
Type and design of study (eg, parallel, crossover, double-blind, open, superiority, noninferiority).Blinding measures taken to minimize bias (eg, "single-blind; subjects receive blinded study medication").

A single arm, multicenter, open-label, prospective study. Requirements for run-in or washout of medication. Those who have been administered one of the following drugs within 2 weeks before they start to participate in this study

* Estrogens
* Antiestrogens
* Progesterones
* Steroids
* Oriental medicines

Description of population to be studied (eg, adults with chronic heart failure and ejection fraction below 40% or subjects with uncontrolled, long-term type 2 diabetes).

Children with central precocious puberty

* Inclusion Criteria.

  1. Female children aged '≥ 4 years ~ < 9 years (8 years plus 364 days)
  2. Those who fall under Tanner stage 2 at least (on condition that they started to have breast budding under the age of 8)
  3. Female children who showed pubertal LH response to GnRH stimulation test (peak ≥ 7mIU/mL)
  4. Those whose bone age increased by one year or more compared to their chronological age
  5. Subjects and their guardians who gave written consent to participate in this study
* Exclusion Criteria.

  1. Those whose bone age is 11 years and 6 months or older
  2. Those secreting gonadal or adrenal cortex sex hormones in a non-LH-dependent manner
  3. Those who have anaphylaxis to the IP or synthetic LHRH, or LHRH derivative
  4. Those who have received GnRH analog treatment
  5. Those who require treatment likely to influence the hypothalamic-pituitary-gonadal axis during the study period
  6. Those receiving growth hormone
  7. Those who are suspected of or diagnosed with malignant tumor
  8. Patients with severe renal failure or hepatic failure, whose participation in this study is impossible in the investigator's opinion
  9. Those who have been administered one of the following drugs within 2 weeks before they started to participate in this study, or who are expected to be administered during the study period

     * Estrogens
     * Antiestrogens
     * Progesterones
     * Steroids
     * Oriental medicines
  10. Those who have participated in another clinical study within 90 days from the date when the IP was administered
  11. Those who are found to be ineligible for this study in the investigator's opinion

ELIGIBILITY:
Inclusion Criteria:

1. Female children aged '≥ 4 years ~ < 9 years (8 years plus 364 days)
2. Those who fall under Tanner stage 2 at least (on condition that they started to have breast budding under the age of 8)
3. Female children who showed pubertal LH response to GnRH stimulation test (peak ≥ 7mIU/mL)
4. Those whose bone age increased by one year or more compared to their chronological age
5. Subjects and their guardians who gave written consent to participate in this study

Exclusion Criteria:

1. Those whose bone age is 11 years and 6 months or older
2. Those secreting gonadal or adrenal cortex sex hormones in a non-LH-dependent manner
3. Those who have anaphylaxis to the IP or synthetic LHRH, or LHRH derivative
4. Those who have received GnRH analog treatment
5. Those who require treatment likely to influence the hypothalamic-pituitary-gonadal axis during the study period
6. Those receiving growth hormone
7. Those who are suspected of or diagnosed with malignant tumor
8. Patients with severe renal failure or hepatic failure, whose participation in this study is impossible in the investigator's opinion
9. Those who have been administered one of the following drugs within 2 weeks before they started to participate in this study, or who are expected to be administered during the study period

   * Estrogens
   * Antiestrogens
   * Progesterones
   * Steroids
   * Oriental medicines
10. Those who have participated in another clinical study within 90 days from the date when the IP was administered
11. Those who are found to be ineligible for this study in the investigator's opinion

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage(%) of subjects with inhibition of LH response (peak <3mIU/mL) | at 24 weeks
  Percentage(%) of subjects with inhibition of LH response (peak <3mIU/mL) maintained upon GnRH stimulation test at 12, 24, and 48 weeks

SECONDARY OUTCOMES:
LH peak/FSH ratio maintained to be <1 upon | at 12, 24, and 48 weeks
  Percentage(%) of subjects with a LH peak/FSH ratio maintained to be <1 upon GnRH stimulation test at 12, 24, and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Soon Hwang, MD, PhD, Principal Investigator — Ajoun university hospital
Locations (1):
- Hwang, Jin Soon, Suwon, South Korea